CLINICAL TRIAL: NCT04624776
Title: Steroid Treatment as Anti-inflammatory and Neuroprotective Agent Following Out-of-Hospital Cardiac Arrest. A Randomized Trial
Brief Title: Steroid Treatment After Resuscitated Out-of-Hospital Cardiac Arrest
Acronym: STEROHCA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christian Hassager (Other)
Responsible Party: Sponsor-Investigator, Christian Hassager, Professor, MD, DMSc, FESC, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT: 2020-000855-11
Record Dates: First submitted 2020-10-12; First posted 2020-11-12 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Cardiac Arrest; Cardiac Arrest With Successful Resuscitation; Post Cardiac Arrest Syndrome; Systemic Inflammatory Response Syndrome; Neurological Injury
Keywords: OHCA; PCAS; Inflammation; Neuroprotection; Methylprednisolone; Solu-Medrol
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest; Post-Cardiac Arrest Syndrome; Systemic Inflammatory Response Syndrome; Trauma, Nervous System; Inflammation | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, 1:1 randomized, multicenter, double-blind, placebo-controlled clinical trial. A minimum of 120 unconscious OHCA patients will be randomized 1:1 after 5 minutes of sustained ROSC to an infusion of 250 mg (4 mL) methylprednisolone in the pre-hospital setting. The methylprednisolone will be given as a bolus infusion of 1 x 250 mg (1 x 4 mL) over a period of 5 minutes. Patients allocated to placebo will receive 4 mL of isotonic saline (NaCl 0.9%).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone (Active Comparator): A five minutes bolus infusion of 250 mg (4 mL) methylprednisolone to inhibit inflammatory and neurological damage following resuscitated out-of-hospital cardiac arrest. The infusion of methylprednisolone will be given following five minutes of sustainable ROSC in the prehospital setting.
  Interventions: Drug: Methylprednisolone
- Isotonic saline (Placebo Comparator): A bolus infusion of 4 mL isotonic saline (NaCl 0.9%).
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Methylprednisolone — A dosis of 250 mg methylprednisolone is suspended in isotonic saline to a total volume of 4 mL prior to infusion.
  Other Names: Solu-Medrol
  Arms: Methylprednisolone
Drug: Isotonic saline — A bolus infusion of 4 mL isotonic saline (NaCl 0.9%).
  Other Names: Placebo
  Arms: Isotonic saline

SUMMARY:
Comatose patients resuscitated from Out-of-Hospital Cardiac Arrest (OHCA) often develop a complicated systemic inflammatory response and have a poor prognosis with neurological damage being the most common cause of death. This study will investigate the anti-inflammatory and neuroprotective effect of early treatment with the glucocorticoid methylprednisolone measured by interleukin-6 and neuron-specific enolase levels in resuscitated comatose OHCA-patients.

DETAILED DESCRIPTION:
BACKGROUND:

Each year approximately 5400 individuals suffer from Out-of-Hospital Cardiac Arrest (OHCA) in Denmark and despite an improved prognosis 30-day mortality is around 90%. For OHCA patients resuscitated successfully and admitted to an Intensive Care Unit (ICU) the 30-day mortality remains higher than 50% due to a complicated systemic response, referred to as the Post Cardiac Arrest Syndrome (PCAS). PCAS consists of four interacting components: 1) ischemic/reperfusion brain injury, 2) myocardial dysfunction, 3) a systemic inflammatory response and 4) persistent stress from the triggering cause of the cardiac arrest, e.g. acute myocardial infarction. PCAS progresses during the first 1-2 days following resuscitated cardiac arrest, and the treatment aims to reduce neurologic injury by cooling the patient to 33-36° C, circulatory support with vasopressors, inotropics or mechanical devices as well as identification and treatment of reversible causes to the cardiac arrest, e.g. acute revascularization of an AMI.

Several studies have shown that the systemic inflammatory response is associated with a high risk of poor outcome following OHCA. Inflammatory markers associated with poor outcome include interleukin (IL) 6, high sensitivity C-reactive protein (hsCRP), leucocytes, IL-1b, IL-10, IL-13, tumor necrosis factor alpha (TNF-alpha) and procalcitonin. Despite of this, there is no specific treatment that addresses this complicated and life-threatening systemic response, and guidelines remain inconclusive in this field.

Anoxic irreversible brain injury remains the leading cause of death following resuscitated OHCA. The complex mechanism is one of the components in the PCAS and is thought to develop due to neuron apoptosis and reperfusion/ischemic injury. Further, the biomarker neuron-specific enolase (NSE) is correlated to neuron damage in the blood stream and has a strong predictive value for poor outcome following OHCA. Inhibiting the causes of the systemic inflammatory response and thereby potentially the brain injury in the very early stages following resuscitation from OHCA may therefore be key to optimizing post-cardiac arrest care.

Following resuscitated OHCA, the function of the adrenal gland is compromised due to global ischemia and reduced levels of the hormone steroid, glucocorticoid, are produced. Glucocorticoid has an important role in several physiologic processes including an anti-inflammatory systemic response. As a result, resuscitated cardiac arrest patients are affected by a severe inflammatory response, while the natural defense mechanism of the body to modulate inflammation is suppressed. Systemic treatment with steroids serves as an anti-inflammatory mediator and counteracts acute microcirculation injury and free radical formation, resulting in diminished vasodilation and reduction of edema, e.g. brain edema. Two small studies have shown signs of improved survival and neurologic outcome among patients who was given injections with glucocorticoids after in-hospital cardiac arrest. The incidence of adverse events was not higher in patients receiving glucocorticoids. Long-term treatment with glucocorticoids is associated with a series of side effects, whereas short-term treatment only has a few side effects. Systemic treatment with glucocorticoids could therefore be an important and safe factor in the treatment of resuscitated cardiac arrest patients that could potentially improve survival and neurological outcome.

Methylprednisolone and other glucocorticoids are used in pulse doses (>250 mg prednisolone equivalent a day) in various acute immunologically mediated conditions/diseases such as organ transplantation to prevent organ rejection and certain rheumatic diseases with acute deterioration. All these conditions are associated with a severe inflammatory response, as seen in PCAS, and therefore methylprednisolone doses as high as 30 mg/kg (equivalent of 2.1 g for a person weighing 70 kg) are used in pulse therapy to obtain an adequate response and effect. Further, the advantage of pulse dose glucocorticoid treatment is better efficacy, but also a decrease in side effects due to a reduced need for longer lasting therapy exceeding days or weeks. The literature reports of possible cardiovascular side effects as bradycardia and arrhythmias associated to infusion of pulse doses of methylprednisolone/glucocorticoids if given within a short period of time, but the evidence is limited and not well supported. The Danish summary of product characteristics recommends an initial infusion of Solu-Medrol to be administered over a period of at least five minutes.

Based on the above knowledge the intervention in this study is 250 mg of methylprednisolone administered intravenously as a bolus infusion over five minutes.

In summary, following resuscitated OHCA, PCAS, a severe and life-threatening condition, is often developed. PCAS is associated with increased mortality and poor neurological outcome. Inhibition of this inflammatory response may have an important, yet relatively unknown, role in post-cardiac arrest care.

HYPOTHESIS:

Bolus infusion of 250 mg methylprednisolone in the pre-hospital setting will inhibit the systemic inflammatory response and minimize the degree of neurological injury in comatose, resuscitated Out-of-Hospital Cardiac Arrest (OHCA) patients.

SAMPLE SIZE:

The trial is powered at the co-primary endpoint. The investigators chose a priori to power the trial at the 'weakest' of the two endpoints, ensuring a sufficient power for both endpoints. As the investigators were not able to find data regarding the effect of methylprednisolone on IL-6 levels or NSE levels from OHCA admission, the trial was powered towards a single measurement drawn 48 hours after admission. In 171 patients from the investigators institution the mean (logarithmically transformed to approximate normal distribution) IL-6 level after 48 hours from admission was 4.19±1.27 (unpublished data). The investigators assumed that methylprednisolone would reduce the IL-6 level by 20%. With an α-level of 0.025, the trial would achieve a power of 0.90 if 112 patients were included. The mean (logarithmically transformed to approximate normal distribution) NSE level after 48 hours was 3.21±0.96 after 48 hours from admission (unpublished data). The investigators assumed that methylprednisolone would reduce the NSE level by 20%. With an α-level of 0.025, the trial would achieve a power of 0.90 if 114 patients were included. The investigators aimed to include 120 patients, to adjust for missingness due to withdrawn consent. Further, since a proportion of the patients were expected to die before complete assessment of the co-primary endpoint (i.e. blood sampling at 72 hours), randomization of patients will continue until a total of 120 patients have survived to blood sampling at 72 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. OHCA of presumed cardiac cause
3. Unconsciousness (GCS ≤8) upon pre-hospital randomization
4. Sustained ROSC for at least 5 minutes
5. Randomization and start of study medicine infusion within 30 minutes of sustained ROSC.

Exclusion Criteria:

1. Advanced life support termination-of-resuscitation exclusion criteria
2. Asystole as primary ECG rhythm
3. Women of childbearing capacity
4. Known therapy limitation
5. Known allergy to methylprednisolone
6. Known pre-arrest modified Rankin Scale (mRS) score of 4-5
7. Temperature upon randomization <30° C
8. >30 minutes to sustained ROSC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Concentration of IL-6 | Daily measurements from admission to 72 hours after admission
  Interleukin 6 (ng/L)
Concentration of NSE | Daily measurements from admission to 72 hours after admission
  Neuron-specific-enolase (ng/L)

SECONDARY OUTCOMES:
Markers of inflammation, biomarkers | Daily measurements the first three days following admission
  High sensitivity C-reactive protein (hsCRP, mg/L) and plasma cytokine levels exemplified by IL-6 (ng/L)
Markers of inflammation, cell count | Daily measurements the first three days following admission
  Leucocyte- and differential count (thousand cells/µL)
Markers of kidney and hepatic injury | Daily measurements the first three days following admission
  Creatinine, ALAT, ASAT, BF and bilirubin (all in mg/L)
Marker of the coagulation system, biomarker | Plasma fibrinogen the first three days from admission
  Plasma fibrinogen (mg/L)
Marker of the coagulation system, functional analysis | Thromboelastography at admission and at 48 hours
  Thromboelastography (TEG, measured in minutes)
Hemodynamics, Swan-Ganz catheter | Daily Swan-Ganz catheter measurements the first five days from admission
  Measurements on Swan-Ganz catheter (CVP, PAP, PCWP - all in mmHg)
Hemodynamics, arterial blood gasses (Lactate) | Arterial blood gasses bihourly the first 36 hours
  Arterial blood gasses (Lactate in mmol/L)
Hemodynamics, arterial blood gasses | Arterial blood gasses bihourly the first 36 hours
  Arterial blood gasses (PaO2 and PaCO2 in kPa)
Neuroprotection, biomarkers | Biomarkers the first three days from admission
  Biomarkers TAU, NFL, NFM, NFH and GFAP (all in mmol/L)
Cardiac protection, biomarkers | Biomarkers the first three days from admission
  TnT, TnI and CKMB (all in mmol/L).
Clinical endpoint, survival | 180 days following discharge
  Survival (yes/no, register based data from "The Medical Register of Births and Deaths" in Denmark)
Clinical endpoint, neurological outcome by mRS score | After five days of admission and at 30- and 180- days following discharge
  Neurological outcome (modified Rankin Scale score, 0-6 symptom scale with higher scores indicating more severe symptoms)
Safety, adverse events | From admission till 7 days following admission
  Cumulated incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hassager, MD, DMSc, Principal Investigator — Department of Cardiology, The Heart Center, Rigshospitalet, Copenhagen, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Gentofte Hospital, Gentofte Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sasson C, Rogers MA, Dahl J, Kellermann AL. Predictors of survival from out-of-hospital cardiac arrest: a systematic review and meta-analysis. Circ Cardiovasc Qual Outcomes. 2010 Jan;3(1):63-81. doi: 10.1161/CIRCOUTCOMES.109.889576. Epub 2009 Nov 10. PMID 20123673
- [Background] Soholm H, Wachtell K, Nielsen SL, Bro-Jeppesen J, Pedersen F, Wanscher M, Boesgaard S, Moller JE, Hassager C, Kjaergaard J. Tertiary centres have improved survival compared to other hospitals in the Copenhagen area after out-of-hospital cardiac arrest. Resuscitation. 2013 Feb;84(2):162-7. doi: 10.1016/j.resuscitation.2012.06.029. Epub 2012 Jul 13. PMID 22796541
- [Background] Neumar RW, Nolan JP, Adrie C, Aibiki M, Berg RA, Bottiger BW, Callaway C, Clark RS, Geocadin RG, Jauch EC, Kern KB, Laurent I, Longstreth WT Jr, Merchant RM, Morley P, Morrison LJ, Nadkarni V, Peberdy MA, Rivers EP, Rodriguez-Nunez A, Sellke FW, Spaulding C, Sunde K, Vanden Hoek T. Post-cardiac arrest syndrome: epidemiology, pathophysiology, treatment, and prognostication. A consensus statement from the International Liaison Committee on Resuscitation (American Heart Association, Australian and New Zealand Council on Resuscitation, European Resuscitation Council, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Asia, and the Resuscitation Council of Southern Africa); the American Heart Association Emergency Cardiovascular Care Committee; the Council on Cardiovascular Surgery and Anesthesia; the Council on Cardiopulmonary, Perioperative, and Critical Care; the Council on Clinical Cardiology; and the Stroke Council. Circulation. 2008 Dec 2;118(23):2452-83. doi: 10.1161/CIRCULATIONAHA.108.190652. Epub 2008 Oct 23. No abstract available. PMID 18948368
- [Background] Stub D, Bernard S, Duffy SJ, Kaye DM. Post cardiac arrest syndrome: a review of therapeutic strategies. Circulation. 2011 Apr 5;123(13):1428-35. doi: 10.1161/CIRCULATIONAHA.110.988725. No abstract available. PMID 21464058
- [Background] Callaway CW, Donnino MW, Fink EL, Geocadin RG, Golan E, Kern KB, Leary M, Meurer WJ, Peberdy MA, Thompson TM, Zimmerman JL. Part 8: Post-Cardiac Arrest Care: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S465-82. doi: 10.1161/CIR.0000000000000262. No abstract available. PMID 26472996
- [Background] Peberdy MA, Andersen LW, Abbate A, Thacker LR, Gaieski D, Abella BS, Grossestreuer AV, Rittenberger JC, Clore J, Ornato J, Cocchi MN, Callaway C, Donnino M; National Post Arrest Research Consortium (NPARC) Investigators. Inflammatory markers following resuscitation from out-of-hospital cardiac arrest-A prospective multicenter observational study. Resuscitation. 2016 Jun;103:117-124. doi: 10.1016/j.resuscitation.2016.01.006. Epub 2016 Jan 27. PMID 26826561
- [Background] Vaahersalo J, Skrifvars MB, Pulkki K, Stridsberg M, Rosjo H, Hovilehto S, Tiainen M, Varpula T, Pettila V, Ruokonen E; FINNRESUSCI Laboratory Study Group. Admission interleukin-6 is associated with post resuscitation organ dysfunction and predicts long-term neurological outcome after out-of-hospital ventricular fibrillation. Resuscitation. 2014 Nov;85(11):1573-9. doi: 10.1016/j.resuscitation.2014.08.036. Epub 2014 Sep 17. PMID 25238742
- [Background] Bro-Jeppesen J, Kjaergaard J, Stammet P, Wise MP, Hovdenes J, Aneman A, Horn J, Devaux Y, Erlinge D, Gasche Y, Wanscher M, Cronberg T, Friberg H, Wetterslev J, Pellis T, Kuiper M, Nielsen N, Hassager C; TTM-Trial Investigators. Predictive value of interleukin-6 in post-cardiac arrest patients treated with targeted temperature management at 33 degrees C or 36 degrees C. Resuscitation. 2016 Jan;98:1-8. doi: 10.1016/j.resuscitation.2015.10.009. Epub 2015 Oct 23. PMID 26525271
- [Background] Bro-Jeppesen J, Kjaergaard J, Wanscher M, Nielsen N, Friberg H, Bjerre M, Hassager C. Systemic Inflammatory Response and Potential Prognostic Implications After Out-of-Hospital Cardiac Arrest: A Substudy of the Target Temperature Management Trial. Crit Care Med. 2015 Jun;43(6):1223-32. doi: 10.1097/CCM.0000000000000937. PMID 25756419
- [Background] Fries M, Kunz D, Gressner AM, Rossaint R, Kuhlen R. Procalcitonin serum levels after out-of-hospital cardiac arrest. Resuscitation. 2003 Oct;59(1):105-9. doi: 10.1016/s0300-9572(03)00164-3. PMID 14580740
- [Background] Laver S, Farrow C, Turner D, Nolan J. Mode of death after admission to an intensive care unit following cardiac arrest. Intensive Care Med. 2004 Nov;30(11):2126-8. doi: 10.1007/s00134-004-2425-z. Epub 2004 Sep 9. PMID 15365608
- [Background] Dragancea I, Rundgren M, Englund E, Friberg H, Cronberg T. The influence of induced hypothermia and delayed prognostication on the mode of death after cardiac arrest. Resuscitation. 2013 Mar;84(3):337-42. doi: 10.1016/j.resuscitation.2012.09.015. Epub 2012 Sep 20. PMID 23000363
- [Background] Schneider A, Bottiger BW, Popp E. Cerebral resuscitation after cardiocirculatory arrest. Anesth Analg. 2009 Mar;108(3):971-9. doi: 10.1213/ane.0b013e318193ca99. PMID 19224811
- [Background] Stammet P, Collignon O, Hassager C, Wise MP, Hovdenes J, Aneman A, Horn J, Devaux Y, Erlinge D, Kjaergaard J, Gasche Y, Wanscher M, Cronberg T, Friberg H, Wetterslev J, Pellis T, Kuiper M, Gilson G, Nielsen N; TTM-Trial Investigators. Neuron-Specific Enolase as a Predictor of Death or Poor Neurological Outcome After Out-of-Hospital Cardiac Arrest and Targeted Temperature Management at 33 degrees C and 36 degrees C. J Am Coll Cardiol. 2015 May 19;65(19):2104-14. doi: 10.1016/j.jacc.2015.03.538. PMID 25975474
- [Background] Wiberg S, Hassager C, Schmidt H, Thomsen JH, Frydland M, Lindholm MG, Hofsten DE, Engstrom T, Kober L, Moller JE, Kjaergaard J. Neuroprotective Effects of the Glucagon-Like Peptide-1 Analog Exenatide After Out-of-Hospital Cardiac Arrest: A Randomized Controlled Trial. Circulation. 2016 Dec 20;134(25):2115-2124. doi: 10.1161/CIRCULATIONAHA.116.024088. Epub 2016 Nov 12. PMID 27838646
- [Background] Schultz CH, Rivers EP, Feldkamp CS, Goad EG, Smithline HA, Martin GB, Fath JJ, Wortsman J, Nowak RM. A characterization of hypothalamic-pituitary-adrenal axis function during and after human cardiac arrest. Crit Care Med. 1993 Sep;21(9):1339-47. doi: 10.1097/00003246-199309000-00018. PMID 8396524
- [Background] Hekimian G, Baugnon T, Thuong M, Monchi M, Dabbane H, Jaby D, Rhaoui A, Laurent I, Moret G, Fraisse F, Adrie C. Cortisol levels and adrenal reserve after successful cardiac arrest resuscitation. Shock. 2004 Aug;22(2):116-9. doi: 10.1097/01.shk.0000132489.79498.c7. PMID 15257083
- [Background] Barnes PJ. Anti-inflammatory actions of glucocorticoids: molecular mechanisms. Clin Sci (Lond). 1998 Jun;94(6):557-72. doi: 10.1042/cs0940557. PMID 9854452
- [Background] Barnes PJ. Molecular mechanisms and cellular effects of glucocorticosteroids. Immunol Allergy Clin North Am. 2005 Aug;25(3):451-68. doi: 10.1016/j.iac.2005.05.003. PMID 16054537
- [Background] Dietrich J, Rao K, Pastorino S, Kesari S. Corticosteroids in brain cancer patients: benefits and pitfalls. Expert Rev Clin Pharmacol. 2011 Mar;4(2):233-42. doi: 10.1586/ecp.11.1. PMID 21666852
- [Background] Varvarousi G, Stefaniotou A, Varvaroussis D, Xanthos T. Glucocorticoids as an emerging pharmacologic agent for cardiopulmonary resuscitation. Cardiovasc Drugs Ther. 2014 Oct;28(5):477-88. doi: 10.1007/s10557-014-6547-4. PMID 25163464
- [Background] Mentzelopoulos SD, Zakynthinos SG, Tzoufi M, Katsios N, Papastylianou A, Gkisioti S, Stathopoulos A, Kollintza A, Stamataki E, Roussos C. Vasopressin, epinephrine, and corticosteroids for in-hospital cardiac arrest. Arch Intern Med. 2009 Jan 12;169(1):15-24. doi: 10.1001/archinternmed.2008.509. PMID 19139319
- [Background] Mentzelopoulos SD, Malachias S, Chamos C, Konstantopoulos D, Ntaidou T, Papastylianou A, Kolliantzaki I, Theodoridi M, Ischaki H, Makris D, Zakynthinos E, Zintzaras E, Sourlas S, Aloizos S, Zakynthinos SG. Vasopressin, steroids, and epinephrine and neurologically favorable survival after in-hospital cardiac arrest: a randomized clinical trial. JAMA. 2013 Jul 17;310(3):270-9. doi: 10.1001/jama.2013.7832. PMID 23860985
- [Background] Caplan A, Fett N, Rosenbach M, Werth VP, Micheletti RG. Prevention and management of glucocorticoid-induced side effects: A comprehensive review: A review of glucocorticoid pharmacology and bone health. J Am Acad Dermatol. 2017 Jan;76(1):1-9. doi: 10.1016/j.jaad.2016.01.062. PMID 27986132
- [Background] Sinha A, Bagga A. Pulse steroid therapy. Indian J Pediatr. 2008 Oct;75(10):1057-66. doi: 10.1007/s12098-008-0210-7. Epub 2008 Nov 21. PMID 19023530
- [Background] Buttgereit F, da Silva JA, Boers M, Burmester GR, Cutolo M, Jacobs J, Kirwan J, Kohler L, Van Riel P, Vischer T, Bijlsma JW. Standardised nomenclature for glucocorticoid dosages and glucocorticoid treatment regimens: current questions and tentative answers in rheumatology. Ann Rheum Dis. 2002 Aug;61(8):718-22. doi: 10.1136/ard.61.8.718. PMID 12117678
- [Background] Jacobs JW, Geenen R, Evers AW, van Jaarsveld CH, Kraaimaat FW, Bijlsma JW. Short term effects of corticosteroid pulse treatment on disease activity and the wellbeing of patients with active rheumatoid arthritis. Ann Rheum Dis. 2001 Jan;60(1):61-4. doi: 10.1136/ard.60.1.61. PMID 11114284
- [Background] Langford CA. Management of systemic vasculitis. Best Pract Res Clin Rheumatol. 2001 Jun;15(2):281-97. doi: 10.1053/berh.2001.0144. PMID 11469822
- [Background] Vasheghani-Farahani A, Sahraian MA, Darabi L, Aghsaie A, Minagar A. Incidence of various cardiac arrhythmias and conduction disturbances due to high dose intravenous methylprednisolone in patients with multiple sclerosis. J Neurol Sci. 2011 Oct 15;309(1-2):75-8. doi: 10.1016/j.jns.2011.07.018. Epub 2011 Aug 9. PMID 21831398
- [Background] Altunbas G, Sucu M, Zengin O. Ventricular repolarization disturbances after high dose intravenous methylprednisolone Theraphy. J Electrocardiol. 2018 Jan-Feb;51(1):140-144. doi: 10.1016/j.jelectrocard.2017.07.017. Epub 2017 Aug 1. PMID 28912075
- [Background] Morrison LJ, Visentin LM, Kiss A, Theriault R, Eby D, Vermeulen M, Sherbino J, Verbeek PR; TOR Investigators. Validation of a rule for termination of resuscitation in out-of-hospital cardiac arrest. N Engl J Med. 2006 Aug 3;355(5):478-87. doi: 10.1056/NEJMoa052620. PMID 16885551
- [Background] Morrison LJ, Verbeek PR, Vermeulen MJ, Kiss A, Allan KS, Nesbitt L, Stiell I. Derivation and evaluation of a termination of resuscitation clinical prediction rule for advanced life support providers. Resuscitation. 2007 Aug;74(2):266-75. doi: 10.1016/j.resuscitation.2007.01.009. Epub 2007 Mar 23. PMID 17383072
- [Derived] Obling LER, Beske RP, Meyer MAS, Grand J, Wiberg S, Damm-Hejmdal A, Bjerre M, Frikke-Schmidt R, Folke F, Moller JE, Kjaergaard J, Hassager C. Inflammatory response after prehospital high-dose glucocorticoid to patients resuscitated from out-of-hospital cardiac arrest: A sub-study of the STEROHCA trial. Resuscitation. 2024 Sep;202:110340. doi: 10.1016/j.resuscitation.2024.110340. Epub 2024 Jul 31. PMID 39094677
- [Derived] Obling LER, Beske RP, Meyer MAS, Grand J, Wiberg S, Mohr T, Damm-Hejmdal A, Forman JL, Frikke-Schmidt R, Folke F, Moller JE, Kjaergaard J, Hassager C. Effect of prehospital high-dose glucocorticoid on hemodynamics in patients resuscitated from out-of-hospital cardiac arrest: a sub-study of the STEROHCA trial. Crit Care. 2024 Jan 22;28(1):28. doi: 10.1186/s13054-024-04808-3. PMID 38254130
- [Derived] Obling LER, Beske RP, Meyer MAS, Grand J, Wiberg S, Nyholm B, Josiassen J, Sondergaard FT, Mohr T, Damm-Hejmdal A, Bjerre M, Frikke-Schmidt R, Folke F, Moller JE, Kjaergaard J, Hassager C. Prehospital high-dose methylprednisolone in resuscitated out-of-hospital cardiac arrest patients (STEROHCA): a randomized clinical trial. Intensive Care Med. 2023 Dec;49(12):1467-1478. doi: 10.1007/s00134-023-07247-w. Epub 2023 Nov 9. PMID 37943300
- [Derived] Obling LER, Beske RP, Wiberg S, Folke F, Moeller JE, Kjaergaard J, Hassager C. Steroid treatment as anti-inflammatory and neuroprotective agent following out-of-hospital cardiac arrest: a randomized clinical trial. Trials. 2022 Nov 22;23(1):952. doi: 10.1186/s13063-022-06838-0. PMID 36414975